CLINICAL TRIAL: NCT02737969
Title: Use of Transesophageal Echocardiography/Angiography Fusion Software Prototype for Structural Heart Disease Procedures
Brief Title: TEE/Angio Fusion Study
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-00048
Record Dates: First submitted 2016-03-24; First posted 2016-04-14 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Structural Heart Disease
Keywords: Transesophageal Echocardiography/angiography (TEE/Angio)
MeSH Terms: interventions — Echocardiography, Transesophageal; Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TEE/Angio fusion software: Patients planned to undergo a transcatheter-based structural heart disease procedure that utilizes TEE and fluoroscopic guidance
  Interventions: Device: Transesophageal Echocardiography/angiography (TEE/Angio)

INTERVENTIONS:
Device: Transesophageal Echocardiography/angiography (TEE/Angio) — The TEE probe will be inserted into the patient's esophagus, after anesthetic induction or conscious sedation is administered, and removed after the completion of the procedure. Once the TEE probe is placed, the interventional cardiologist will acquire 2 fluoroscopic images with the TEE probe. These images will be used to co-register the ultrasound and fluoroscopy systems. As part of routine care, TEE and fluoroscopy images will be acquired throughout the procedure for clinical purposes. As new fluoroscopy images are acquired, the prototype software will automatically track the location of the TEE probe. When the echocardiographer has an image of a cardiac structure of interest, he may use the prototype software to place landmarks.
  The echocardiographer may then press a button to have the landmarks displayed on the fluoroscopy image that is only visible on an assist monitor and will not interfere with the standard fluoroscopy imaging monitor.

SUMMARY:
This is a pilot study of patients undergoing structural heart disease procedures that utilize TEE and fluoroscopic guidance at the New York University (NYU) Langone Medical Center. Patients in this study will undergo their procedure utilizing the TEE/Angio fusion software prototype. This protocol is primarily intended to ascertain the potential utility of the software prototype in the study population and to provide data and feedback to improve the workflow and algorithms of the prototype. As such, a primary outcome variable and statistical analysis plan have not been identified. However, procedural time, measures of radiation exposure (dose area product, total radiation dose, fluoroscopy time), degree of residual valvular regurgitation or paravalvular regurgitation as applicable, and complications will be recorded.

DETAILED DESCRIPTION:
This study is for patients planned to undergo a transcatheter-based structural heart disease procedure that utilizes TEE and fluoroscopic guidance at the NYU Langone Medical Center. It will evaluate the utility and workflow of the transesophageal echocardiography/angiography (TEE/Angio) fusion software prototype to provide visualization of anatomic landmarks and guidance during structural heart disease procedures.

The purpose of this study is to evaluate software (TEE/Angio fusion) that merges images from two standard procedures (ultrasound and x-ray) used to look at the heart during a procedure for structural heart disease. Typically, these 2-dimensional images are viewed separately, requiring the operator to mentally merge the two images together while deciding if he/she is in the correct location for the treatment strategy. TEE/Angio fusion is designed to make a single 3-dimensional image of the heart in real-time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be more than 18 years of age
* Subjects must have a plan to undergo a transcatheter-based structural heart disease procedure that utilize TEE and fluoroscopic guidance

Exclusion Criteria:

* Subjects with a known contraindication for insertion of the TEE probe (e.g. history of esophageal stricture, scleroderma, etc.), which will be ascertained by a non-invasive imaging specialist (contraindications are routinely assessed in the course of the preoperative workup)Subjects who have a known contraindication for insertion of the TEE probe (e.g. history of esophageal stricture, scleroderma, etc.), which will be ascertained by a non-invasive imaging specialist (contraindications are routinely assessed in the course of the preoperative workup)
* Pregnant
* Participating in a competing study
* Unable or do not provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned to undergo a transcatheter-based structural heart disease procedure that utilizes TEE and fluoroscopic guidance at the NYU Langone Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Procedural Time' | One day
Dose Area Product of Radiation Exposure | One day
  Once the TEE probe is placed, the interventional cardiologist will acquire 2 fluoroscopic images with the 'tee probe in view, at least 30 degrees apart. These 2 images will be used to co-register the ultrasound and fluoroscopy systems. The document entitled, "NSR_EchoXrayFusion", this adds a negligible amount of radiation exposure (0.0006%).
Degree of residual valvular or paravalvular regurgitation | One day
Total Radiation Dose | One Day
Fluoroscopy Time | One Day

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Williams, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States